CLINICAL TRIAL: NCT00731744
Title: Generation of Dendritic Cell Precursors From Cord Blood Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chien-Nan Lee, National Taiwan Unviersity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200706003R
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Normal Full-Term Deliveries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Normal full-term deliveries — Normal full-term deliveries by standard procedures according to institutional guidelines

SUMMARY:
There is a growing interest in generating dendritic cells (DCs) for using as vaccines. Several cytokines, especially stem cell factor (SCF) and FLT3-ligand (FL), have been identified as essential to produce large numbers of myeloid precursors and even to increase DC yield obtained by the action of granulocyte-macrophage colony-stimulating factor (GM-CSF) and tumor necrosis factor alpha (TNF-α). However, there are few studies on the effect of the early-acting cytokines, commonly used to expand CD34+ progenitor cells, on DC generation.

We have established a serious of functional analysis of maturated or immaturated DCs including surface markers screening or cytokine production. Here, we design this two-year project to evaluate the possible methodology in the generation of CD14+CD1a- and CD14- CD1a+ myeloid DC precursors from CD34+ cells. In the first year of the project, we will set up the standard protocol to generate DC precursors from cord blood stem cells. In the first step, we will isolate CD34+ cells from cord blood and amplify these cells. Purity of the CD34+ cell populations obtained will be greater than 90%. In the next step, these primary cultures of CD34+ cells will treat with early-acting cytokines such as GM-CSF and IL-4 to further induction into dendritic cells. Functional analysis of dendritic cells would be performed in this stage. In the second year of the project, we will further evaluate the induction of DCs by CD34+ stem cells could be affected by combination of mesenchymal stromal cells. These results of this research with CD34+-based DCs induction provide the basis for materials to develop the DC-based vaccine against viral and fungal infections, and might be a powerful tool in anti-tumor immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Normal full-term deliveries

Exclusion Criteria:

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
None, we isolate stem cells from cord blood. | from CS operation to close

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan